CLINICAL TRIAL: NCT06913660
Title: A Smartphone Game to Increase Engagement in Care Among African Adolescents Living With HIV
Brief Title: ALHIV Smartphone Game Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate Winskell, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002974; 5R33MH124200-04 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-04-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hiv; AIDS; Adolescent Behavior; Treatment Compliance; Treatment Adherence; Reproductive Behavior; Sexual Behavior
Keywords: HIV; Smartphone Game
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Adolescent Behavior; Patient Compliance; Treatment Adherence and Compliance; Reproductive Behavior; Sexual Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A cluster-randomized feasibility study, that involves clinic-level randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention is an Android smartphone-based interactive narrative-driven game called MyGoals.
  Participants will be instructed to play the game for at least 30 minutes for 5 days per week for the first 6 weeks and as desired thereafter.
  Interventions: Behavioral: MyGoals
- Control Arm (Active Comparator): Control-arm participants will receive the current standard of care offered at their CCC (i.e. HIV care management support and counselling received at the CCC).
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: MyGoals — A smartphone game for ALHIV aged 15-21 yrs
  MyGoals includes 3 components:
  1. A role-playing narrative in which all players make decisions for male and female characters navigating scenarios from adolescence and early adulthood.
  2. A series of mini-games to reinforce knowledge, skills and related self-efficacy, explored in the narrative.
  3. A metanarrative component, My Story, where players will create an avatar and set personal goals.
  Arms: Intervention Arm
Behavioral: Standard of care — A minimum standard of care package will be identified prior to identification and recruitment of CCCs to ensure a comparable and adequate level of care is being offered to all control participants, since implementation of the range of support and care strategies recommended by the Kenya Ministry of Health differs by clinic.
  Other Names: Standard of care package
  Arms: Control Arm

SUMMARY:
This is a cluster-randomized controlled trial that aims to conduct comprehensive feasibility testing of a smartphone game in a sample of 120 adolescents living with HIV (ALHIV) ages 15-21 in Kisumu, Kenya, to determine whether the game influences behavioral mediators of engagement in care and sexual risk avoidance and reduction (including knowledge, attitudes, behavioral intentions, and self-efficacy).

DETAILED DESCRIPTION:
This is a cluster-randomized feasibility study that will involve clinic-level randomization of 120 ALHIV participants (12 from each of 10 clinical centers). Participants will either use the intervention (a smartphone game) or continue standard treatment and support for HIV. Participants will complete 5 surveys about behaviors, attitudes, knowledge, and self-efficacy relating to engagement in care, ART adherence, and sexual and reproductive health. They will also have blood drawn 3 times to measure their HIV viral load. Intervention-arm participants will also complete app experience surveys. A sample of intervention-arm participants will be invited to provide feedback on their experience in interviews (n=10) and/or focus groups (n=30).

ELIGIBILITY:
Adolescents, male and female, aged 15-21 in Kisumu County (n=120)

Inclusion criteria:

* Aged 15-21 at time of recruitment
* Diagnosed with HIV and aware of HIV status
* Initiated ART at least 6 months prior
* Accesses HIV-related care at intervention arm CCC
* VL above 50 copies/ml at last test, with last test conducted within 12 months prior to recruitment date

Exclusion criteria

* Does not have basic literacy in English (Grade 3-4 on the Flesch-Kincaid Reading Scale)
* Sibling to an adolescent already enrolled in study
* Sibling to adolescent that participated in formative research
* Participant in formative research to inform study
* Participant in any Tumaini game activities
* Enrolled in boarding school
* Last recorded viral load test >12 months prior to recruitment date

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Knowledge measures will be assessed via Yes/No//I do not know survey questions and will address ART (antiretroviral therapy), HIV, sexually transmitted infections (STIs), pregnancy, and condoms. Answers to knowledge questions will be coded as 0 or 1, with higher scores indicating more accurate knowledge. Total possible score range is 0-14. A positive value for the change from baseline score will indicate an increase in knowledge from the baseline assessment.
Change in attitudes | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Attitudes will be assessed via Likert survey questions relating to HIV stigma, condoms, sex, and gender. Attitudes items will be scored on a 0-1 scale, with higher scores indicating more desirable attitudes. Total possible score range is 0-14. A positive value for the change from baseline score will indicate an increase in desirable attitudes.
Change in behavioral intentions | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Behavioral intention will be assessed via Likert survey questions. The measure will address intention to avoid risk and to engage in health protective behaviors. Behavioral intention items will be scored on a 0-1 scale with higher scores indicating more intention to partake in health protective behaviors and a positive value for the change from baseline score indicating an increase in intention to engage in health protective behaviors. Total possible score range is 0-9.
Change in self-efficacy | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Self-efficacy will be assessed via a Likert scale, and focus on self-efficacy for condom use; to communicate with a partner about protected sex; to adhere to medication; to fully engage in care and to disclose their HIV status. Self-efficacy will be scored on a 0-1 scale with higher scores indicating stronger self-efficacy. A positive value for the change from baseline score will indicate an increase in self-efficacy since the baseline assessment. Total possible score range is 0-23.
Change in game acceptability | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Acceptability will be assessed among intervention-arm participants via Likert scale questions. Acceptability will be scored on a 0-1 scale with higher scores indicating higher acceptability. Total possible score range is 0-12, with higher score correlating with better study outcome.
Change in game immersion | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Immersion will be assessed among intervention-arm participants via Likert scale questions and focus on identification, transportation, and immersion. Immersion items will be scored on a 0-1 scale with higher scores indicating stronger immersion. Total possible score range is 0-18. Higher score correlates with better study outcome.
Change in game continued use | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Continued use of the intervention over the course of the study will be assessed among intervention-arm participants via both self-report survey questions and analysis of paradata. Survey items will assess self-reported use of the game in hours at each follow-up study timepoint. Paradata analysis will calculate time in hours spent on the app for each intervention-arm participant.
Change in game demand | Baseline, 9 months post-intervention
  Demand for ongoing access to the intervention following study endline will be assessed among intervention-arm participants via Likert scale questions. Demand items will be scored on a 0-1 scale with higher scores indicating stronger demand. Total possible score range is 0-2, and higher score correlates with better study outcome.
Change in game safety | Baseline, 6 weeks, 3 months, 6 months and 9 months post-intervention
  Participants' perceived safety while in possession of the phone and app will be assess among intervention-arm participants via Likert scale questions. These will focus on physical safety as well as comfort with having an HIV-related app on the study phone. Safety items will be scored on a 0-1 scale with higher scores indicating higher perceived safety. Total possible score range is 0-4, and higher score correlates with better study outcome.

SECONDARY OUTCOMES:
Change in viral load (VL) from baseline | Baseline, mid-point (around 4 months post-intervention), and endline (9 months post-intervention)
  VL will be assessed as "undetectable" (<50 copies/ml) or "detectable".
Change in attendance at scheduled clinic visits | Baseline, 9 months post-intervention
  Participant medical records (MR) will be used to review attendance.
Change in Retention in care | Baseline, 9 months post-intervention
  Retention in care will be assessed as "disengaged" (has missed the last scheduled appointment and over half of all scheduled appointment within the previous study period) or "engaged".

CONTACTS AND LOCATIONS:
Overall Officials: Kate Winskell, PhD, Principal Investigator — Emory University
Locations (1):
- KEMRI Clinical Research Centre, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT06913660/ICF_000.pdf